CLINICAL TRIAL: NCT05733299
Title: Automating Patient Inhaler Technique When Using Pressurised Metered Dose Inhalers: Testing the Functionality and Impact of the Aflo™ Digital Respiratory Management Platform in a Randomised Controlled Trial.
Brief Title: Aflo™ Device Trial
Acronym: AFLO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ulster (Other)
Collaborators: Northern Ireland Clinical Research Service (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22.WM.0278
Record Dates: First submitted 2023-01-20; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Asthma; Asthma in Children
Keywords: asthma; asthma control; respiratory management platform; medical device; inhaler technique
MeSH Terms: conditions — Asthma | interventions — Standard of Care

STUDY DESIGN:
Masking Description: Independent allocation, no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator)
  Interventions: Other: Standard care
- aflo™ digital respiratory management platform with standard care (Experimental): The new aflo™ digital respiratory management platform will provide automated inhaler technique direction, with real time quantitative personalised feedback on inhaler technique and timing.
  Interventions: Device: aflo™ digital respiratory management platform; Other: Standard care

INTERVENTIONS:
Device: aflo™ digital respiratory management platform — medical device, user app, clinician portal, data analytics hub
  Arms: aflo™ digital respiratory management platform with standard care
Other: Standard care — Health service standard care will be continued

SUMMARY:
This randomised, prospective, controlled parallel study aims to evaluate the role and potential of the aflo™ digital platform for improving asthma control, inhalation technique and adherence in patients who use metred dose inhalers (MDI). The study will recruit 104 patients with uncontrolled asthma in the North-West of Northern Ireland. Fifty two patients will remain on standard care over 24-weeks and 52 will combine standard care with the aflo™ platform. The data collected over a 24-week period will be used to determine 1. whether the aflo™platform improves inhalation technique and user adherence to prescribed medication and 2. Lead to better asthma control and reduced symptoms as measured by the Asthma Control Test (ACT). During the study clinicians will be able to remotely monitor and review user analytics via a clinical dashboard. ACT measurements will be recorded at start and end of study. The study aims to test the functionality and impact of automated inhaler technique with real-time feedback, adherence prompts and air quality data sharing for patients who use metered dose inhalers (MDI) using the newly developed aflo™ digital respiratory management platform.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed as suitable for inclusion by their General Practitioner or asthma nurse.
* Access to WiFi and a smart phone (Android or apple phone with latest version -2) and knowledge of / carer support with using a smartphone.
* For children (parent/ carer must register and provide smart phone access)
* Aged > 5 years (with carer/ parental consent if < 17 years old)
* Smart phone user/ willing to use (or parent/ carer) and have access to and knowledge of working a smart phone and WIFI / 4G
* Currently prescribed an inhaled reliever +/- preventer medication via pressurised
* Metered Dose Inhaler (MDI) short acting beta2 agonist (SABA), inhaled corticosteroid (ICS) ICS / long acting beta2 agonist (LABA) MDI +/- spacer
* Adherence/ symptom control issues with medication (as identified by excess use of SABA/ healthcare personnel visits/ calls/ emergency department visit/ hospital admission
* Those who understand written and spoken English

Exclusion Criteria:

* < 5 years old
* Other major respiratory illness or significant concurrent disease that might prevent completion of the study

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-02-06 (Estimated); Primary Completion 2024-02-05 (Estimated); Study Completion 2024-02-05 (Estimated)

PRIMARY OUTCOMES:
Inhaler Proficiency checklist Score (IPS) | Change over 24 weeks
  Inhalation score 0-7 (higher the score the greater the proficiency)

SECONDARY OUTCOMES:
Asthma control | Change over 24 weeks
  Asthma Control Test (ACT) (0-25 with a score <20: uncontrolled; 20-24: reasonably well controlled; 25: controlled)
Medication usage | Change over 24 weeks
  Usage of asthma medication: increased usage of 'preventer' inhaler and decreased use of salbutamol/' reliever' inhaler
Health impairment in asthma patients | Change over 24 weeks
  Measured by St George's Respiratory Questionnaire (SGRQ).(0: best health; 100: worse health)
Lung function | Change over 24 weeks
  Lung volume / capacity measured by a spirometer
Lung function | Change over 24 weeks
  Lung rates of flow measured by a spirometer
Lung function | Change over 24 weeks
  Lung gas exchange measured by a spirometer
Inflammation | Change over 24 weeks
  Blood immunoglobulin E (IgE) (microarray)
Inflammation | Change over 24 weeks
  Blood eosinophils (Sysmex full blood count)
Exhaled breath nitric oxide (FeNO) | Change over 24 weeks
  Measured by a FeNO monitoring system
Asthma health and symptoms questionnaire | Change over 24 weeks
  Number of hospital visits, number of attacks (the higher number the more negative the outcome).

OTHER OUTCOMES:
Patient satisfaction | At 24 weeks
  Evaluation of device (4-point scale; higher score the more satisfied)
Device feedback | Baseline, 12 weeks and 24 weeks
  Functionality of device (4-point scale; higher score the more satisfied)
Qualitative feedback | Baseline, 12 weeks and 24 weeks
  Unstructured open-ended feedback

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Human Intervention Studies Unit, Coleraine, N.Ireland
  - Health Hub Professionals, Londonderry, N.Ireland

IPD SHARING:
Plan to Share IPD: No
Commercially sensitive